CLINICAL TRIAL: NCT02348112
Title: A Post-Market Evaluation of the Altis® Single Incision Sling System Versus Transobturator or Retropubic Mesh Sling in the Treatment of Female Stress Urinary Incontinence
Brief Title: Altis® 522 Trial - Treatment of Female Stress Urinary Incontinence
Status: Completed | Type: Observational
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: SU020
Record Dates: First submitted 2015-01-16; First posted 2015-01-28 (Estimated); Results first posted 2023-11-21 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: Stress Urinary Incontinence
Keywords: stress urinary incontinence; Altis 522; urinary incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress; Urinary Incontinence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Altis arm: Subjects will have an Altis sling placed to treat stress urinary incontinence.
  Interventions: Device: Altis Single Incision Sling
- Comparator arm: Subjects will have a transobturator or retropubic sling placed to treat stress urinary incontinence.
  Interventions: Device: Transobturator or Retropubic Sling

INTERVENTIONS:
Device: Altis Single Incision Sling — Altis is a minimally invasive, adjustable incontinence sling that is placed through a single incision in the vaginal wall and anchored inside the body. The sling has an integrated tensioning system eliminating the need for additional skin exits.
  Groups: Altis arm
Device: Transobturator or Retropubic Sling — Both transobturator and retropubic slings are a hammock-like mesh placed underneath the urethra to provide support. A single incision is made in the vaginal wall and two incisions in the abdomen. Tensioning of the sling is achieved by pulling the sling through the abdominal incisions.
  Groups: Comparator arm

SUMMARY:
The aim of this postmarket study is to compare the safety and effectiveness of the Altis Single Incision Sling (SIS) to an FDA cleared transobturator and/or retropubic sling through 36 months.

DETAILED DESCRIPTION:
This study is a prospective, post-market, multi-center, cohort assessment comparing Altis SIS (n=178) and transobturator and/or retropubic slings (n=178) in the treatment of stress urinary incontinence at up to 40 U.S. and international sites. Subjects will be followed for a total of 36 months with scheduled visits at 6, 12, 18, 24 and 36 months. The study population will consist of adult female subjects with stress urinary incontinence who are clinically indicated for surgical intervention with a mesh sling.

ELIGIBILITY:
Inclusion Criteria:

* The subject is female and at least 18 years of age.
* The subject is able and willing to complete all procedures and follow-up visits indicated in this protocol.
* The subject has confirmed stress urinary incontinence (SUI) through cough stress test or urodynamics.
* The subject has failed two non-invasive incontinence therapies (such as Kegel exercise, behavior modification, pad use, biofeedback, etc.) for > 6 months.

Exclusion Criteria:

* The subject has an active urogenital infection or active skin infection in region of surgery.
* The subject has confirmed Pelvic Organ Prolapse (POP) of Stage 2 or higher as determined by POP-Q prolapse grading.
* The subject is having a concomitant pelvic floor procedure.
* The subject has incontinence due to neurogenic causes (e.g. multiple sclerosis, spinal cord/brain injury, cerebrovascular accident, detrusor-external sphincter dyssynergia, Parkinson's disease, or similar conditions).
* The subject had a prior surgical stress urinary incontinence (SUI) treatment.
* The subject has undergone radiation or brachy therapy to treat pelvic cancer.
* The subject has urge predominant incontinence by MESA assessment.
* The subject has an atonic bladder or post void residual (PVR) above 100 cc on ≥ 2 occasions.
* The subject is pregnant and/or is planning to get pregnant in the future.
* The subject has a contraindication to the surgical procedure or the product Instructions for Use (IFU).
* The subject is enrolled in a concurrent clinical trial of any treatment (drug or device) that could affect continence function, without the sponsors approval.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be selected from urology or urogynecology specialties.
Sampling Method: Non-Probability Sample
Enrollment: 416 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2021-09 (Actual); Study Completion 2021-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ty Erickson, MD, Principal Investigator — Rosemark WomenCare Specialists
Locations (27):
- United States (26):
  - Stanford University, Stanford, California
  - Pelvic Solutions Center, Denver, Colorado
  - Urology Specialists, LLC, Hialeah, Florida
  - Rosemark Women Care Specialists, Idaho Falls, Idaho
  - Women's Health Advantage, Fort Wayne, Indiana
  - Boston Urogynecology Associates, Cambridge, Massachusetts
  - Baystate Health System, Springfield, Massachusetts
  - Female Pelvic Medicine & Urogynecology, Grand Rapids, Michigan
  - Adult and Pediatric Urology & Urogynecology, Omaha, Nebraska
  - University of Nevada, Las Vegas, Nevada
  - Albany Medical Center, Albany, New York
  - Associated Urologists of North Carolina, Cary, North Carolina
  - Novant Health, Charlotte, North Carolina
  - Carolina Urology Partners, Gastonia, North Carolina
  - FirstHealth Urogynecology, Hamlet, North Carolina
  - Associated Urologists of North Carolina, Raleigh, North Carolina
  - Lyndhurst Clinical Research, Winston-Salem, North Carolina
  - Akron Urogynecology Associates, Akron, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Genesis Healthcare, Zanesville, Ohio
  - University of Oklahoma, Oklahoma City, Oklahoma
  - The Institute for Female Pelvic Medicine and Reconstructive Surgery, Allentown, Pennsylvania
  - Institute of Female Pelvic Medicine & Reconstructive Surgery, North Wales, Pennsylvania
  - Lexington Urology, West Columbia, South Carolina
  - Sanford Health, Sioux Falls, South Dakota
  - The Group for Women, Virginia Beach, Virginia
- CHUS Hopital Fleurimont, Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Erickson T, Gheiler E, Hanson CE, McCrery R, Parekh M, Parva M, Tu LM. Patient Satisfaction and QoL in SUI: Results With Single-Incision or Full-Length Slings. Urogynecology (Phila). 2025 Oct 1;31(10):942-951. doi: 10.1097/SPV.0000000000001586. PMID 39423154
- [Derived] Erickson T, Roovers JP, Gheiler E, Parekh M, Parva M, Hanson C, McCrery R, Tu LM. A Multicenter Prospective Study Evaluating Efficacy and Safety of a Single-incision Sling Procedure for Stress Urinary Incontinence. J Minim Invasive Gynecol. 2021 Jan;28(1):93-99. doi: 10.1016/j.jmig.2020.04.014. Epub 2020 Apr 19. PMID 32320798

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Altis Arm | Comparator Arm
Started | 213 | 203
Completed | 140 | 101
Not Completed | 73 | 102
Not completed — Withdrawal by Subject | 32 | 29
Not completed — Lost to Follow-up | 24 | 20
Not completed — Physician Decision | 17 | 15
Not completed — Site closed due to PI leaving | 0 | 30
Not completed — Sponsor withdrawal | 0 | 7
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) analysis population is all enrolled subjects. A subject is considered enrolled once signed informed consent is obtained.
Groups:
- Total: Total of all reporting groups
Arm/Group | Altis Arm | Comparator Arm | Total
Number analyzed (Participants) | 213 | 203 | 416
Age, Categorical [Count of Participants; unit: Participants] — Population: 2 participants in the Altis arm and 1 participant in the Comparator arm with age unknown.
  Participants
    number analyzed (Participants) | 211 | 202 | 413
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 153 | 155 | 308
    >=65 years | 58 | 47 | 105
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: 2 participants in the Altis arm and 1 participant in the Comparator arm with age unknown.
  years
    number analyzed (Participants) | 211 | 202 | 413
    (all) | 56.4 (11.8) | 53.6 (12.0) | 55.1 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 213 | 203 | 416
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 55 | 25 | 80
  Not Hispanic or Latino | 156 | 177 | 333
  Unknown or Not Reported | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 12 | 15
  White | 205 | 181 | 386
  More than one race | 1 | 3 | 4
  Unknown or Not Reported | 4 | 5 | 9
Region of Enrollment [Number; unit: participants]
  United States | 169 | 203 | 372
  Canada | 44 | 0 | 44
Pad Weight (g) [Mean (Standard Deviation); unit: grams] — Population: 14 participants in the Altis arm and 16 participants in the Comparator arm with pad weight test not done.
  grams
    number analyzed (Participants) | 199 | 187 | 386
    (all) | 88.0 (155.8) | 96.8 (154.7) | 92.3 (155.1)

OUTCOME MEASURES:

1. Primary Outcome: Primary Effectiveness Endpoint
Description: Observed effectiveness, defined as a reduction from baseline in 24 hour pad weight of at least 50% at 6 months.
Time Frame: 6 months
Population: All enrolled subjects (Intent-to-Treat (ITT) analysis population) who have undergone a sling implant attempt for stress urinary incontinence using either Altis SIS or an FDA cleared transobturator or retropubic sling (modified Intent-to-Treat (mITT) analysis population). The mITT analysis population is a subset of the ITT population. The mITT analysis population is the primary analysis population for the assessment of all safety and effectiveness endpoints.
Measure: Count of Participants; unit: Participants
Arm/Group | Altis Arm | Comparator Arm
Number analyzed (Participants) | 167 | 143
Participants | 130 | 119
Statistical Analysis 1: Comparison: Altis Arm vs Comparator Arm; Test type: Non-Inferiority — The number and proportion of subjects experiencing a 50% or greater reduction in pad weight at 6 months were compared, and non-inferiority assessed using a normal approximation test (Z-test) for a difference in binomial proportion. Non-inferiority was considered achieved if the 95% confidence interval for the difference in proportions (Comparator - Altis) was less than 0.15; p = 0.013, Normal approximation test (Z-test); Difference in Proportions = -0.054, 95% CI 2-sided [-0.139 to 0.031]

2. Primary Outcome: Primary Safety Endpoint
Description: Observed device and/or procedure-related serious adverse events through 36 months.
Time Frame: 36 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Altis Arm | Comparator Arm
Number analyzed (Participants) | 184 | 171
Participants | 2 | 4
Statistical Analysis 1: Comparison: Altis Arm vs Comparator Arm; Test type: Non-Inferiority — The number and proportion of subjects experiencing device- and/or procedure-related serious adverse events were tabulated for each study group. Non-inferiority through 36 months was calculated using a normal approximation test (Z-test) for a difference in binomial proportion. Non-inferiority was considered achieved if the lower limit of the 95% confidence interval for the difference in proportions (Comparator - Altis) is greater than -0.10 in the mITT analysis population; p < 0.0001, Normal approximation test (Z-test); Difference in Proportions = 0.013, 95% CI 2-sided [-0.023 to 0.048]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected through 36 months.
Arm/Group | Altis Arm | Comparator Arm
All-Cause Mortality (participants affected / at risk) | 0/184 | 1/171
Serious Adverse Events (participants affected / at risk) | 24/184 | 29/171
Other Adverse Events (participants affected / at risk) | 74/184 | 66/171
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Altis Arm (N=184) | Comparator Arm (N=171)
Bleeding, hematoma or hemorrhage (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Delayed wound healing (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Mesh exposure (extrusion) (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Shortness of breath, chest pain, L jaw/neck pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pelvic / urogenital pain (groin) (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Perforation, bladder (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Urinary retention/obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Abdominal Abscess following appendectomy (Infections and infestations) | 1 (1) | 0 (0)
Acute pancreatitis (Endocrine disorders) | 0 (0) | 1 (1)
Acute renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Adenomyosis (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Appendicitis (Gastrointestinal disorders) | 2 (2) | 1 (1)
Broke left arm (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Broke right arm (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Broken left ankle (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Broken right ankle (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cervical Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Diverticular stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Elective surgery of total prosthesis right knee (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Exacerbation of COPD (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (4)
Femur fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Hydrocephalus (Nervous system disorders) | 1 (1) | 0 (0)
Intra-abdominal abscess (Infections and infestations) | 1 (1) | 0 (0)
Left Carotid Stenosis (Vascular disorders) | 1 (1) | 0 (0)
Left Humerus Fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Metastatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Morbid Obesity (General disorders) | 0 (0) | 1 (1)
Non STEMI myocardial Infarction (Cardiac disorders) | 1 (1) | 0 (0)
Parastomal abscess and cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Paroxysmal Atrial Fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Partial small bowel obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Patient hurt her shoulder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Perianal abscess (Infections and infestations) | 0 (0) | 1 (1)
Pre-Cancerous Cells Removed From Left Breast (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Rectal Bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0)
Retro-sternal pain (Cardiac disorders) | 1 (1) | 0 (0)
Right Elbow fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Right Shoulder Reconstructive Surgery (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Right bimalleolar ankle fracture, fibular fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Right carpal tunnel release surgery (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Small bowel obstruction and fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Thoracic Degenerative Discs (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Total right knee prothesis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Worsening Right knee pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Abdominal tenderness (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abnormal cardiac stress test (Cardiac disorders) | 0 (0) | 1 (1)
Abnormal mammogram (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bilateral knee pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Drug overdose (General disorders) | 0 (0) | 1 (1)
Endometrial cancer (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Increased blood sugars (Endocrine disorders) | 0 (0) | 1 (1)
Left femur fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Medial meniscus tear of right knee (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Ocular migraine (General disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Pulmonary thromboembolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Recurrent gluteus Medius tear (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Right coronary occlusion (Cardiac disorders) | 0 (0) | 1 (1)
Right index finger and thumb injury (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Small bowel obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Spinal cord stimulator (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Total left knee prothesis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Unstable angina / chest pains (Cardiac disorders) | 0 (0) | 1 (1)
Wound necrosis (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Altis Arm (N=184) | Comparator Arm (N=171)
Urinary retention/obstruction (Renal and urinary disorders) | 11 (11) | 3 (3)
Hip pain (Musculoskeletal and connective tissue disorders) | 8 (8) | 2 (2)
Pelvic / urogenital pain (groin) (Musculoskeletal and connective tissue disorders) | 10 (10) | 5 (5)
Nausea (Gastrointestinal disorders) | 5 (5) | 0 (0)
Dyspareunia, de novo (Reproductive system and breast disorders) | 16 (16) | 5 (5)
Leg pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0)
Hip and leg pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Recurrent incontinence (Renal and urinary disorders) | 7 (7) | 12 (12)
Dyspareunia, worsening (Reproductive system and breast disorders) | 3 (3) | 1 (1)
Urgency, worsening (Renal and urinary disorders) | 2 (2) | 14 (15)
Infection (Infections and infestations) | 0 (0) | 2 (2)
Urinary tract infection (Renal and urinary disorders) | 39 (61) | 39 (96)
Urgency, de novo (Renal and urinary disorders) | 5 (5) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 3 (3) | 1 (1)

LIMITATIONS AND CAVEATS:
The strengths of the Altis 522 Study include its large sample size, prospective, multicenter design and use of a wide variety of standardized and validated instruments to collect patient reported outcomes over a 36-month study duration. Potential limitations associated with the study include rates of enrollment, subject attrition rates, and differences in baseline characteristics.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-11-01): https://cdn.clinicaltrials.gov/large-docs/12/NCT02348112/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-08): https://cdn.clinicaltrials.gov/large-docs/12/NCT02348112/SAP_001.pdf